CLINICAL TRIAL: NCT06575686
Title: A Phase 2 Study of Epcoritamab Plus Tazemetostat for Treatment of Relapsed/Refractory Follicular Lymphoma
Brief Title: Epcoritamab and Tazemetostat for the Treatment of Relapsed or Refractory Grade I-IIIa Follicular Lymphoma
Status: Suspended | Phase: Phase 2 | Type: Interventional
Why Stopped: Pending Interim Analysis
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 23820; NCI-2024-06708 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 23820 (Other: City of Hope Medical Center); P30CA033572 (NIH)
Record Dates: First submitted 2024-08-23; First posted 2024-08-28 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Recurrent Grade 1 Follicular Lymphoma; Recurrent Grade 2 Follicular Lymphoma; Recurrent Grade 3a Follicular Lymphoma; Refractory Grade 1 Follicular Lymphoma; Refractory Grade 2 Follicular Lymphoma; Refractory Grade 3a Follicular Lymphoma
MeSH Terms: conditions — Lymphoma, Follicular | interventions — Specimen Handling; Biopsy; Magnetic Resonance Spectroscopy; tazemetostat

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (epcoritamab, tazemetostat) (Experimental): Patients receive tazemetostat PO BID on days 1-28 of each cycle. Patients also receive epcoritamab SC on days 1, 8, 15, and 22 of cycles 2-4 then on day 1 of remaining cycles. Cycles repeat every 28 days for up to 13 cycles in the absence of disease progression or unacceptable toxicity. Patients also undergo collection of blood samples on study and undergo bone marrow biopsy and CT or PET/CT throughout the study.
  Interventions: Procedure: Biospecimen Collection; Procedure: Bone Marrow Biopsy; Procedure: Computed Tomography; Biological: Epcoritamab; Procedure: Positron Emission Tomography; Drug: Tazemetostat

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Bone Marrow Biopsy — Undergo bone marrow biopsy
  Other Names: Biopsy of Bone Marrow; Biopsy, Bone Marrow
Procedure: Computed Tomography — Undergo CT or PET/CT
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; tomography
Biological: Epcoritamab — Given SC
  Other Names: Anti-CD20/CD3 Bispecific Antibody GEN3013; DuoBody-CD3xCD20; Epcoritamab-bysp; Epkinly; GEN 3013; GEN-3013; GEN3013; Tepkinly
Procedure: Positron Emission Tomography — Undergo PET/CT
  Other Names: Medical Imaging, Positron Emission Tomography; PET; PET Scan; Positron emission tomography (procedure); Positron Emission Tomography Scan; Positron-Emission Tomography; proton magnetic resonance spectroscopic imaging; PT
Drug: Tazemetostat — Given PO
  Other Names: E 7438; E-7438; E7438; EPZ 6438; EPZ-6438; EPZ6438

SUMMARY:
This phase II trial tests the safety, side effects and effectiveness of epcoritamab and tazemetostat in treating patients with grade I-IIIa follicular lymphoma that has come back after a period of improvement (relapsed) or that has not responded to previous treatment (refractory). Epcoritamab is a bispecific monoclonal antibody that binds to two different antigens on the surface of cancer cells that may help the body's immune system attack the cancer and may interfere with the ability of the cancer cells to grow and spread. Tazemetostat, a EZH2 inhibitor, may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth. Giving epcoritamab and tazemetostat may be safe, tolerable and/or effective in treating patients with relapsed or refractory grade I-IIIa follicular lymphoma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To assess the safety/tolerability of epcoritamab in combination with tazemetostat in patients with relapsed/refractory follicular lymphoma (FL). (Safety lead-In) II. To evaluate the anti-tumor activity of epcoritamab in combination with tazemetostat in patients with relapsed/refractory FL by complete response rate. (Phase II)

SECONDARY OBJECTIVES:

I. To estimate overall response rate (ORR) duration of response (DOR) of the combination of epcoritamab and tazemetostat.

II. To estimate progression-free survival, and overall survival of the combination of epcoritamab and tazemetostat.

III. To assess the toxicities of the combination of epcoritamab and tazemetostat.

EXPLORATORY OBJECTIVES:

I. To characterize the T-cell population balance in patients treated with epcoritamab and tazemetostat in different compartments (peripheral blood, tumor).

II. To explore correlation between response and presence of EZH2 mutations. III. To evaluate minimal residual disease (MRD) dynamics during treatment and explore the correlation of MRD kinetics with response.

OUTLINE:

Patients receive tazemetostat orally (PO) twice daily (BID) on days 1-28 of each cycle. Patients also receive epcoritamab subcutaneously (SC) on days 1, 8, 15, and 22 of cycles 2-4 then on day 1 of remaining cycles. Cycles repeat every 28 days for up to 13 cycles in the absence of disease progression or unacceptable toxicity. Patients also undergo collection of blood samples on study and undergo bone marrow biopsy and computed tomography (CT) or positron emission tomography (PET)/CT throughout the study.

After completion of study treatment, patients are followed up at 30 and 60 days then for up to 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Documented informed consent of the participant and/or legally authorized representative

  * Assent, when appropriate, will be obtained per institutional guidelines
* Agreement to allow the use of archival tissue from diagnostic tumor biopsies

  * If unavailable, exceptions may be granted with study principal investigator (PI) approval
* Age: ≥ 18 years
* Eastern Cooperative Oncology Group (ECOG) ≤ 2
* Histologically confirmed follicular lymphoma, grades 1-3A
* Relapsed/ refractory disease after at least one line of prior lymphoma therapy
* Radiologically measurable lymphadenopathy (≥ 1.5 cm) or ≥ 1 measurable extranodal lesion (long axis > 1.0 cm) on CT scan or magnetic resonance imaging (MRI)
* Fully recovered from the acute toxic effects (except alopecia) to ≤ grade 1 to prior anti-cancer therapy
* WITHOUT BONE MARROW INVOLVEMENT: Absolute neutrophil count (ANC) ≥ 1,000/mm^3 (NOTE: Growth factor use is allowed to reach ANC)
* WITH BONE MARROW INVOLVEMENT: ANC ≥ 500/mm^3 (NOTE: Growth factor use is allowed to reach ANC)
* WITHOUT BONE MARROW INVOLVEMENT: Platelets ≥ 50,000/mm^3 (NOTE: Platelet transfusions are within 14 days of platelet assessment if thrombocytopenia is secondary to disease involvement)
* WITH BONE MARROW INVOLVEMENT: Platelets ≥ 25,000/mm^3 (NOTE: Platelet transfusions are within 14 days of platelet assessment if thrombocytopenia is secondary to disease involvement)
* Total bilirubin ≤ 2 x upper limit of normal (ULN) (unless has Gilbert's disease or secondary to disease)
* Aspartate aminotransferase (AST) ≤ 2.5 x ULN
* Alanine aminotransferase (ALT) ≤ 2.5 x ULN
* Creatinine clearance of ≥ 45 mL/min per 24 hour urine test or the Cockcroft-Gault formula
* If not receiving anticoagulants: International normalized ratio (INR) OR prothrombin (PT) ≤ 1.5 x ULN; If on anticoagulant therapy: PT must be within therapeutic range of intended use of anticoagulants
* If not receiving anticoagulants: Activated partial thromboplastin time (aPTT) ≤ 1.5 x ULN; If on anticoagulant therapy: aPTT must be within therapeutic range of intended use of anticoagulants
* Fridericia's formula-corrected QT interval (QTcF) ≤ 480 ms (Note: To be performed within 28 days prior to day 1 of protocol therapy)
* If seropositive for HIV, hepatitis C virus (HCV) or hepatitis B virus (HBV), nucleic acid quantitation must be performed. Viral load must be undetectable. HIV-infected patients on effective anti-retroviral therapy with undetectable viral load within 6 months are eligible for this trial
* Meets other institutional and federal requirements for infectious disease titer requirements (Note Infectious disease testing to be performed within 28 days prior to day 1 of protocol therapy)
* Women of childbearing potential (WOCBP): negative serum pregnancy test
* Agreement by females of childbearing potential must agree to either abstain from heterosexual intercourse or to use two effective methods of birth control simultaneously (effective methods described below). The time period for effective contraceptive requirements begins ≥ 28 days prior to initiating tazemetostat and for the course of the study treatment period through at least 6 months after the last dose of tazemetostat, 4 months after the last dose of epcoritamab, or 4 months after the last dose of tocilizumab (if applicable), whichever is longer. Childbearing potential is defined as not being surgically sterilized (men and women) or have not been free from menses for > 1 year (women only). Two effective methods includes one highly effective method and one barrier method.

  * Highly effective methods:

    * Intrauterine device (IUD)
    * Intrauterine hormone-releasing system (IUS)
    * Hormonal (stopping ovulation with two drugs [estrogen and progesterone]: oral, within the vagina, or on/under the skin; stopping ovulation with one drug progesterone-only: oral, injected, or on/under the skin). NOTE: Due to the potential of tazemetostat interference with hormonal contraception methods, use of these method requires that you add a barrier method of contraception (preferably male condom)
    * Bilateral tubal ligation
    * Partner's vasectomy (if medically confirmed there are no live sperm and sole sexual partner)
  * Barrier methods:

    * Male latex or synthetic condom
    * Diaphragm
    * Cervical cap
* Agreement by males to either practice complete abstinence or agree to use a latex or synthetic condom, even with a successful vasectomy (medically confirmed azoospermia), during sexual contact with a female of childbearing potential from first dose of study drug, during study treatment (including during dose interruptions), and for 3 months after study drug discontinuation. NOTE: Male subjects must not donate semen or sperm from first dose of tazemetostat, during study treatment (including during dose interruptions), and for 3 months after discontinuation of tazemetostat

Exclusion Criteria:

* Concurrent enrollment in another therapeutic investigational study
* Prior bispecific antibodies or tazemetostat
* Autologous stem cell transplant within 30 days prior to day 1 of protocol therapy
* Allogeneic stem cell transplant if complicated by active graft versus host disease (GVHD) or if on immunosuppressive agents
* Chemotherapy, radiation therapy, biological therapy, immunotherapy within 21 days or five half-lives (whichever is shorter for non-radiation therapy) prior to day 1 of protocol therapy
* Immunosuppressive agents other than prednisolone 20 mg daily or equivalent
* Major surgery within 4 weeks of first dose of study drug
* Vaccination with live vaccines within 4 weeks of the first dose of study drug
* Strong and moderate CYP3A4 inducers/ inhibitors within 14 days prior to day 1 of protocol therapy
* Current evidence of central nervous system involvement by the lymphoma
* Currently active, clinically significant cardiovascular disease, such as uncontrolled arrhythmia, or NYHA (New York Heart Association) heart failure class III-IV, or a history of myocardial infarction, unstable angina, or acute coronary syndrome within 6 months of screening
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to study agent
* History of active human immunodeficiency virus (HIV) or active with hepatitis C virus (HCV) or hepatitis B virus (HBV)

  * Participants who are positive for hepatitis B core antibody, hepatitis B surface antigen (HBsAg), or hepatitis C antibody must have a negative polymerase chain reaction (PCR) result before enrollment. Those who are PCR positive will be excluded
* Known active severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) infection

  * If a patient has signs/symptoms suggestive of SARS-CoV-2 infection or have had recent known exposure to someone with SARS-CoV-2 infection, the patient must have a negative molecular (e.g., PCR) test, or 2 negative antigen test results at least 24 hours apart, to rule out SARS-CoV-2 infection

    * Note: SARS-CoV-2 diagnostic tests should be applied following local requirements/recommendations
  * Subjects who do not meet SARS-CoV-2 infection eligibility criteria must be screen failed and may only rescreen after they meet the following SARS-CoV-2 infection viral clearance criteria:

    * No signs/symptoms suggestive of active SARS-CoV-2 infection
    * Negative molecular (e.g., PCR) result or 2 negative antigen test results at least 24 hours apart
    * SARS-CoV-2 testing is only required if a patient has signs/symptoms suggestive of SARS-CoV-2 infection or have had recent known exposure to someone with SARS-CoV-2 infection. Patients who fit this description must have a negative molecular (e.g., PCR) test, or 2 negative antigen test results at least 24 hours apart, to rule out SARS-CoV-2 infection
* Clinically significant uncontrolled illness
* Uncontrolled active systemic infection
* Any prior history of myeloid malignancies, including myelodysplastic syndrome (MDS)/acute myeloid leukemia (AML) or myeloproliferative neoplasm (MPN) or any prior history of T lymphoblastic leukemia (T-LBL)/T acute lymphoblastic leukemia (T-ALL) or B acute lymphoblastic leukemia (B-ALL)
* Other active malignancy. Patients with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen are eligible for this trial. Exceptions are:

  * Malignancy treated with curative intent and no known active disease present for ≥ 3 years prior to initiation of therapy on current study
  * Adequately treated non-melanoma skin cancer or lentigo maligna (melanoma in situ) without evidence of disease
  * Adequately treated in situ carcinomas (e.g., breast, cervical, esophageal, etc.) without evidence of disease
  * Asymptomatic prostate cancer managed with "watch and wait" strategy or hormonal therapy
* Inability to take oral medication or have malabsorption syndrome or any other uncontrolled gastrointestinal condition (e.g., nausea, diarrhea, vomiting) that might impair the bioavailability of tazemetostat
* Females only: Pregnant or breastfeeding
* Any other condition that would, in the investigator's judgment, contraindicate the patient's participation in the clinical study due to safety concerns with clinical study procedures
* Prospective participants who, in the opinion of the investigator, may not be able to comply with all study procedures (including compliance issues related to feasibility/logistics)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Estimated)
Dates: Start 2025-03-11 (Actual); Primary Completion 2028-07-16 (Estimated); Study Completion 2028-07-16 (Estimated)

PRIMARY OUTCOMES:
Incidence of unacceptable adverse events (Safety lead-in) | up to first 2 cycles of study treatment
  Observed toxicities will be summarized by type, severity, and attribution. (each cycle is 28 days)
Complete response (CR) rate | Up to 3 years
  CR rate will be defined as a best response of CR according to Lugano criteria before any documented disease progression or any subsequent non-Hodgkin lymphoma (NHL) treatment. CR rate will be estimated along with the 95% exact binomial confidence interval.

SECONDARY OUTCOMES:
Overall response rate (ORR) | Up to 3 years
  ORR will be defined as a best response of CR or partial response (PR) according to Lugano 2016 guidelines on study before any documented disease progression or any subsequent NHL treatment. ORR will be estimated along with the 95% exact binomial confidence interval.
Duration of response (DOR) | From CR or PR to disease progression/relapse or death, up to 3 years
  DOR will be estimated using the product-limit method of Kaplan and Meier along with the Greenwood estimator of standard error, and 95% confidence interval will be constructed based on log-log transformation. Median DOR will be estimated when possible.
Progression-free survival (PFS) | From start of protocol treatment to disease relapse/progression or death, up to 3 years
  PFS will be estimated using the product-limit method of Kaplan and Meier along with the Greenwood estimator of standard error, and 95% confidence interval will be constructed based on log-log transformation. Median PFS will be estimated when possible.
Overall survival (OS) | From start of protocol treatment to death, up to 3 years
  OS will be estimated using the product-limit method of Kaplan and Meier along with the Greenwood estimator of standard error, and 95% confidence interval will be constructed based on log-log transformation. Median OS will be estimated when possible.
Incidence of adverse events | Up to 60 days after last dose of study drug
  Adverse events will be evaluated and graded using Common Terminology Criteria for Adverse Events version 5.0. Cytokine release syndrome and or immune effector cell associated neurotoxicity syndrome will be evaluated using American Society for Transplantation and Cellular Therapy Consensus grading criteria. Observed toxicities will be summarized by type, severity, and attribution.

CONTACTS AND LOCATIONS:
Overall Officials: Swetha Kambhampati, Principal Investigator — City of Hope Medical Center
Locations (2):
- United States (2):
  - City of Hope Medical Center, Duarte, California
  - City of Hope at Irvine Lennar, Irvine, California